CLINICAL TRIAL: NCT03093805
Title: Clinical Effectiveness of Calcipotriene in Acute Graft Versus Host Disease of the Skin: A Pilot Study
Brief Title: Topical Vitamin D in Acute Graft Versus Host Disease of the Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-6739
Record Dates: First submitted 2017-03-23; First posted 2017-03-28 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Graft Vs Host Disease
Keywords: Hematopoietic Stem Cell Transplant; Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — calcipotriene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Calcipotriene (Experimental): Patients will apply Calcipotriene cream 2 times per day for 7 days.
  Interventions: Dietary Supplement: Calcipotriene

INTERVENTIONS:
Dietary Supplement: Calcipotriene — Topical vitamin D cream will be applied to affected areas of the skin.
  Other Names: Dovonex

SUMMARY:
The purpose of this study is to evaluate the efficacy of Calcipotriene cream. This is a synthetic vitamin D3 derivative for topical use. It is used to treat grade 1-3 acute skin graft versus host disease (GVHD) in hematopoietic stem cell transplant (HSCT) recipients. Calcipotriene will be used as the exclusive topical therapy in addition to standard of care GVHD treatment prescribed for the study subject by the primary physician.

DETAILED DESCRIPTION:
Acute skin GVHD affects about one third of pediatric and adult transplant recipients. Chronic GVHD (cGVHD) affects 40-60% of adult patients who have undergone allogeneic HSCT. It is a major cause of non-relapse mortality and morbidity. Systemic prednisone is the first-line treatment for cGVHD; however, about one-half of all patients do not respond to this initial therapy, and there is no standard second-line therapy. Immunosuppressive therapy used for treatment of GVHD brings significant risk of infection, poorly affecting clinical outcomes.

Vitamin D affects immunoregulation, fibroblast proliferation, collagen synthesis and endothelial cell function, and the investigators hypothesize that topical vitamin D application will have a positive effect on acute and chronic skin GVHD. The investigators hypothesize that topical vitamin D cream may restore normal cell function and decrease the use of steroid creams in acute GVHD of the skin.

ELIGIBILITY:
Inclusion Criteria:

* HSCT recipients with acute Grade I through III GVHD based on Glucksberg criteria. Recipients of multiple transplants are still eligible to participate in this research study.
* Each study subject is to have calcium and vitamin D level prior to starting study, if not obtained within 30 days of beginning treatment.

Exclusion Criteria:

* Patient with active cellulitis at the start of the treatment.
* Patients with hypercalcemia or vitamin D levels above 100 μg/L.
* Patients with known allergy to any of the topical therapy components.
* Patients who have received previous treatment with topical vitamin D cream.

Ages: 3 Months to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
GVHD Grade | 7 days
  Change in GVHD grade over 7 days. GVHD grade based on Glucksberg criteria

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Wallace, DO, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No